CLINICAL TRIAL: NCT05565716
Title: Supporting Self-Management of Healthy Behaviors Among People With Diabetes, Kidney Disease, and Hypertension (SMART-HABITS-4-Health): A Pilot Trial of a Blood Pressure Monitoring Intervention Leveraging Social Incentives and Gamification
Brief Title: Supporting Self-Management of Healthy Behaviors in Diabetes, Kidney Disease, and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 851515; K23DK118198 (NIH)
Record Dates: First submitted 2022-07-05; First posted 2022-10-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Renal Insufficiency, Chronic; Hypertension; Diabetes
Keywords: social incentive; gamification; mHealth; self-management
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Support Person (Experimental): A support person not in the study will receive the participant's weekly blood pressure performance details and will contact them at least on a weekly basis to encourage continued blood pressure monitoring. Prior to randomization, the participant will select a preference between a support person that is close to them (e.g., friend or family member) or a support person who is provided by the study, a Peer Mentor.
  Interventions: Other: Support Person
- Social Norms (Experimental): In this arm, participants will be texted reports of blood pressure performance statistics of the other participants in the study and also receive weekly feedback about how their blood pressure information compares to others in the study. Participants in this arm will have access to a leaderboard that displays this information.
  Interventions: Other: Social Norms

INTERVENTIONS:
Other: Support Person — Prior to randomization, participants will select their preference of the type of support person if they are assigned to this arm 1) a person they have close relationship with, or 2) a Peer Mentor, an individual who has successfully monitored their blood pressure at home using the study's equipment and also has diabetes, kidney disease, and high blood pressure. The Peer Mentor works with the research study team.
  This will be provided with the same weekly blood pressure feedback that the participants will receive. The support person is encouraged to reach out to the participant at least weekly.
  Other Names: Social Support; Peer Mentor
  Arms: Support Person
Other: Social Norms — Participants will receive weekly text messages that includes their individualize blood pressure performance statistics, included frequency of blood pressure monitoring and average blood pressure, and compare it to goals provided at the beginning of the study, as well as the week prior. Participants will also has access to a leaderboard that displays blood pressure performance information all people in the study in an anonymous fashion.
  Other Names: comparative information; normative feedback
  Arms: Social Norms

SUMMARY:
The planned intervention, entitled, Supporting Self-Management of Health Behaviors to Optimize Health (SMART-HABITS for Health), aims to provide support for patients with chronic kidney disease (CKD), hypertension and diabetes by providing text messages delivered as motivational reminders and support to encourage blood pressure self-monitoring through goal setting, customized task prompts via text message and feedback, leveraging social connections, and use of a gamification design.

DETAILED DESCRIPTION:
The pilot trial is designed to study the feasibility of a smartphone-based behavioral intervention in a two groups of participants diagnosed with chronic kidney disease (CKD), diabetes, and hypertension. The patients will be identified for eligibility by screening the scheduled for follow up appointments in the Penn renal CKD clinics. Patients will be prospectively enrolled after informed consent. Participants will be prospectively enrolled and will be randomized to participate into one of two arms.

* Arm 1: Social Support - the participant's performance shared with an identified personal support person, such as a friend or a family member or a Peer Mentor; the support person is encouraged to support the participant on at least a weekly basis. Prior to randomization, each participant will select their preference of a personal support personal or a Peer Mentor. A Peer Mentor is a person also with CKD, HTN, and diabetes who has successfully incorporated regular blood pressure monitoring into their lives.
* Arm 2: Social norms -Participants will have access to a leaderboard of all people in the study that shows blood pressure performance information (frequency and control). They will also receive weekly feedback regarding their personal blood pressure performance, compare to their individualized goals and from the preceding week.

All participants will receive text message reminders sent to prompt blood pressure self-monitoring at least 5 times per week, transmit the blood pressure readings to the secure Way to Health server via Omron Connect app. If a blood pressure reading is not received within 5 hours, another reminder will be sent. Automated text message feedback will be sent after the blood pressur reading is recorded with a tailored message regarding any further required actions based upon the BP readings obtained. Any participant with a single systolic blood pressure reading 200mmHg or two consecutive systolic blood pressure readings 180 mmHg or diastolic blood pressure readings 110 mmHg will be contacted immediately by an MD (Dr. Schrauben) for assessment (including evaluation for symptoms of hypertensive emergency) and referral to the emergency department, if indicated. Please see full text message algorithm (attached protocol). Any participant will undergo re-engagement protocol for low participation.

To further support behavior engagement, there is a gamification element to the design:

* At the beginning of each week (Monday), all participants will receive 70 points (10 points for each day of the week). If participants do not send a BP each day, they will lose 10 points. The goal is to check blood pressure at least 4 days per week.
* All participants will start the study at the second of five levels. At week's end (Sunday), if a participant has ≥40 points, their average systolic blood pressure was in their individualized controlled goal, or their average BP declined from the week prior, they will move up a level to acknowledge goal attainment and improvement, and if not, they will drop a level.
* If a participant reaches the 4th level out of five, they will receive a digital trophy. At study's end, if they accumulate ≥5 trophies, they will receive a mug.
* If a participant reaches the 5th level, they will receive a digital medal. At study's end, if they accumulate ≥4 medals, they will receive a tote bag.
* Each week, participants will receive 50 points to leverage "fresh-start effect"

At the end of the study, each participant will be invited to participate in focus groups for additional feedback on their experience.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic kidney disease (any stage), hypertension, diabetes
* followed at University of Pennsylvania nephrology practice
* aged 18 years or over. -
* own a smart device (smartphone or tablet) capable of connecting to the internet and has Bluetooth enabled technology
* able to comprehend English.
* a mean blood pressure reading of <180/100 mmHg in person study visit
* able and willing to provide informed consent

Exclusion Criteria:

* inability to provide consent or read or speak English
* inability to self-monitor (e.g., diagnosis of dementia, cognitive impairment, physically unable to set up BP cuff and machine)
* already participating in another blood pressure study or intervention trial
* vulnerable populations, living in a long-term care or rehabilitation institution,
* if likely to have their care transferred to another facility outside participating clinic areas during the course of the study
* planning to travel or live consecutively out of the country for more than one month
* mean blood pressure reading of >180/100 mmHg at in person study visit
* hypertension not managed by the nephrologist in Penn Medicine
* any other reason they do not expect to be able to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: Adoption | Collected throughout study (8 weeks)
  Composite outcome determined by participant retention rate, total number of assessments performed by participants over complete study period; Good adoption will be determined by greater than or equal to 70 percent of those retained in the study, and greater than or equal to 70 percent of those enrolled who actually used SMART-HABITS-4-Health at least one time as measured by data usage statistics.
Feasibility: Adherence | Collected throughout study (8 weeks)
  Determined by the number of blood pressure assessments performed divided by the number of assessments recommended. Good adherence will be determined by greater than or equal to 70 percent performed out of the recommended.
Feasibility: Acceptability of SMART-HABITS-4-Health | collected at 4 weeks
  Determined through satisfactory ratings system usability scale survey (score above 68)
Feasibility: Acceptability of SMART-HABITS-4-Health | collected at 8 weeks
  Determined through satisfactory ratings system usability scale survey (score above 68)
Feasibility: Acceptability of SMART-HABITS-4-Health | Collected with 12 weeks of study completion
  Determined by inductive qualitative analysis from semi-structured interviews with study participants after the end of the pilot study. There is no a priori set up codes or scales to assess this outcome as it is purely a qualitative outcome.

SECONDARY OUTCOMES:
Social Incentive Effectiveness | 8 weeks
  Determined by comparing the mean change in baseline BP (the baseline visit BP) to mean BP after 4 and 8 weeks in both arms.
CKD Knowledge | 8 weeks
  Determined by change in enrollment survey and end of study survey scores on responses regarding CKD knowledge using the 28-question Kidney Knowledge Survey (KiKS). The survey score is defined as the sum of the correct responses to each survey question divided by the total number of questions, total score range (0-1). Higher scores indicate better knowledge.
Self-Efficacy | 8 weeks
  Determined by change in enrollment survey and end of study survey scores on responses regarding self-efficacy using the Self-Efficacy for Managing Chronic Disease 6-Item Scale. Answers range from 1 = not at all confident to 10= totally confident, with summary scores indicating higher self-efficacy.
Chronic Disease Self-Management | 8 weeks
  Determined by change in enrollment survey and end of study survey scores on responses regarding self-management using the Partners in Health Scale for Chronic Condition Self-Management (11 items). Answers range from 0=very good to 8= very poor, with higher summary scores indicating better self-management.
Disease Related Quality of Life | 8 weeks
  Determined by change in enrollment survey and end of survey scores on responses regarding disease-related quality of life using the Kidney Disease and Quality of Life 36-item survey (KDQOL-36). Scores are reported separately for each of the five KDQOL-36 subscales and as a summary score. Scores are split into tertiles (thirds) based on the mean of the study population: More than one standard deviation above the mean is the "above average" tertile; The mean +/- one standard deviation is "average" tertile; More than one standard deviation below the mean is the "below average" tertile. Higher scores (both sub-scales and summary) indicate better quality of life.
Maintenance | 8 weeks
  Determined by the usage of SMART-HABITS-4-Health. Good maintenance will be determined by at least one access to the SMART-HABITS-4-Health portal or one BP monitor each week.
Implementation Issues | 8 weeks
  Qualitative reports describing adaptions that were made to the SMART-HABITS program in response to participant feedback, including descriptions of alterations that were made to the schedule of reminders and messaging content. Participant feedback data will be collected with field notes from verbal conversations and textual data from email and text messages.
Reach | 8 weeks
  Determined by the comparison of the sex frequency (percentage) of the enrolled participants compared to sex frequency of general population with chronic kidney disease, diabetes, and with hypertension in the United States.
Reach | 8 weeks
  Determined by the comparison of race (Black, White other) frequency (percentage) of the enrolled participants compared to the race frequencies of the general population with chronic kidney disease, diabetes, and with hypertension in the United States.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schrauben, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No